CLINICAL TRIAL: NCT01454219
Title: Measurement of Glycaemic Responses of Bakery and Confectionery Products
Acronym: GIFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Life Sciences Ltd. (Other)
Collaborators: Fazer (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: GIFA
Record Dates: First submitted 2011-10-14; First posted 2011-10-18 (Estimated); Last update posted 2012-02-15 (Estimated); Status verified 2011-11

CONDITIONS: Healthy

INTERVENTIONS:
Other: Bakery and confectionary products — Control product: Glucose solution, Test products: 11 bakery and confectionary products

SUMMARY:
This study aims to determine the glycemic index, glycemic load and insulin index of eleven Fazer bakery and confectionary products.

ELIGIBILITY:
Inclusion Criteria:

* voluntarily given written consent for participation in research
* healthy man or women, age between 18 ang 65 years
* regular eating
* Body Mass Index 18,5 - 24,9 kg/m2

Exclusion Criteria:

* diabetes
* gastrointestinal diseases
* hepatic, kidney, pancreas or thyroid disease or disorder
* arthritis
* pregnancy or breast feeding
* smoking
* allergy
* severe diseases
* blood donation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Glycemic index (GI)
  The 2 hours glycemic responses to bakery and confectionery products (the incremental area under the glucose response curve, IAUC).

SECONDARY OUTCOMES:
Insulin index (II)
  The 2 hours insulinemic responses to bakery and confectionery products (the incremental area under the insulin response curve, IAUC).
Glycemic load (GL)

CONTACTS AND LOCATIONS:
Overall Officials: Päivi Cheney, MD, Principal Investigator; Tiina Suutari, M.Sc., Study Director — Clinical Life Sciences Ltd.
Locations (1):
- Clinical Life Sciences Ltd, Kajaani, Finland